CLINICAL TRIAL: NCT00904072
Title: Integrated a Novel Clinical Decision Support System (CDSS) in a Computerized Physician Order Entry System
Brief Title: Integrated Novel Clinical Decision Support System (CDSS) in a Computerized Physician Order Entry System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Fe-Lin Lin Wu/Associate Professor, Grauduate Institute of Clinical Pharmacy, College of medicine, National Taiwan university, Grauduate Institute of Clinical Pharmacy
Other Study IDs: 20080306OR
Record Dates: First submitted 2009-05-17; First posted 2009-05-19 (Estimated); Last update posted 2009-05-19 (Estimated); Status verified 2009-05

CONDITIONS: Evaluate the Impact of the CDSS
Keywords: CDSS; prescribing error; prescribing errors influenced by CDSS; CPOE

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- accepted: The suggestions provided by the CDSS which were accepted by the physicians.
- denied: The suggestions provided by the CDSS which were denied by the physicians.

SUMMARY:
The purpose of this study is to understand the impact of CDSS by knowing the prescribers actions to the CDSS, also the influence of prescribing error announced by pharmacists.

DETAILED DESCRIPTION:
1. To assess the sensitivity of the CDSS which could identify some specific prescribing errors (ex: duplication of drugs, dosage that exceed the maximum dose,prescribes drugs that have drug-drug interactions).
2. To identify what kind of drugs are most likely to cause duplication use by the physicians, and what kind of drugs are most likely to exceed the maximum dosage, also to know what kind of drugs are most likely to cause drug-drug interaction that physicians encounter during prescribing.
3. To evaluate the percentage of physician acceptance of the prescribing errors identify by the CDSS.
4. What's the impact of CDSS on pharmacist announced prescribing error.

ELIGIBILITY:
Inclusion Criteria:

* The prescriptions which induced the alert windows pop out.

Exclusion Criteria:

* The prescriptions which not induced the alert windows pop out.

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The prescriptions which induced the alert windows pop out.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2009-02

CONTACTS AND LOCATIONS:
Overall Officials: Fe-Lin Lin Wu, Associate Professor, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital Taipei, Taiwan, Taipei, Taiwan